CLINICAL TRIAL: NCT01955382
Title: Effect of Oral Activated Charcoal on Parasite Clearance Rates in Response to Intravenous Artesunate in Malian Children With Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Evaluation of Oral Activated Charcoal on Antimalarial Drug's Ability to Kill Parasites in Malian Children With Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 999913209; 13-I-N209 (Other: NIAID IRB); NCT01955382 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2013-09-28; First posted 2013-10-07 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Malaria; Severe Malaria
Keywords: Parasite Clearance Rate; Parasite Half Life; Actidose Aqua; Severe Malaria
MeSH Terms: conditions — Malaria; Anthrax | interventions — Charcoal; Artesunate; Injections; Amodiaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AS + oAC (Experimental): All children will receive Artesunate (AS) 2.4 mg/kg IV at 0 and 12 h, 24 h, and 48 h. Children in the AS+oAC group will be given weight-based doses of oAC (Actidose Aqua) (Table 1) at 0, 6, 12, and 18 h. All children will then receive amodiaquine.
  Interventions: Drug: Actidose Aqua; Drug: Artesunate; Drug: Amodiaquine
- AS only (water) (Placebo Comparator): Children in the AS only group will receive a weight-based volume of clean water (Bottled Water) to drink rather than the oAC.
  Interventions: Drug: Artesunate; Drug: Amodiaquine

INTERVENTIONS:
Drug: Actidose Aqua — Actidose Aqua (oAC) (Paddock Laboratories is sold over the counter in the United States in bottles containing 25 g/120 mL (NDC # 0574-0121-04) or 50 g/240 mL (NDC # 0574-0121-08). oAC is stable at room temperature.
  Other Names: Oral activated charcoal
  Arms: AS + oAC
Drug: Artesunate — Artesunate (AS) obtained from Guilin Pharma (Shanghai), the only pharmaceutical company GMP pre-qualified by the WHO. The product artesunate for injection + 5% sodium carbonate inj + 0.9% sodium chloride inj will be delivered in vials of 30 mg and 60- mg vials, respectively, and will be dosed at 2.4 mg/kg as recommended for SM treatment by the WHO
  Other Names: Artesunate for injection
Drug: Amodiaquine — Amodiaquine obtained from Pfizer (Dakar), is provided as 200-mg tablets or syrup (50 10 mg/mL), and will be provided as age-based doses per the manufacturer's directions.
  Other Names: Camoquine

SUMMARY:
Background:

- Malaria is caused by small parasites carried by some mosquitoes. People can get malaria if an infected mosquito bites them. Malaria destroys red blood cells. Most malaria is mild, but some children develop severe malaria, which kills about 660,000 people annually. About 9 in 10 who die of malaria are Sub-Saharan African children, most under 5 years old. Scientists can save many lives if they find out how to prevent or relieve severe malaria.

Objective:

- To know if a common medicine called activated charcoal can reduce severe malaria symptoms.

Eligibility:

- Children 2 to 11 years old with mild malaria who live in Kenieroba, Mali.

Design:

* For the first 2 days and nights, participants will stay in the hospital.
* They will have their medical history taken, and a physical exam.
* Blood will be drawn from a thin tube inserted in their hand or forearm. This will be done 3 times overall. A drop of blood will be taken from a finger prick 12 times overall.
* An antimalarial drug will be injected into the tube in the arm 4 times. Each time the drug is given, participants will drink a small cup of either water or activated charcoal.
* For the following 3 days, participants will take an antimalarial pill.
* On day 7, participants will visit the hospital. A drop of blood from a finger prick will be tested for malaria parasites.

DETAILED DESCRIPTION:
While the incidence of Plasmodium falciparum malaria declines (1) the proportion of cases with severe malaria (SM) may increase (2). The mortality associated with SM in endemic countries remains high despite the use of artesunate (AS) (3). Safe, cheap, and effective adjunct therapies preventing the development of, or reducing the mortality from, SM could have considerable and rapid public health impact. We discovered that oral administration of activated charcoal (oAC), a safe treatment for acute poisoning (4), protects mice from experimental cerebral malaria and demonstrated in a randomized controlled trial (RCT) in African adults that oAC is safe and does not interfere with the pharmacokinetics of AS (5). Here, we propose the next step to evaluate the efficacy of adjunct treatment with oAC in Malian children and to explore its mode of action. Before testing adjunct treatment with oAC in children with SM, we will perform an open-label RCT in children with uncomplicated malaria (UM) to demonstrate non-inferiority of intravenous (IV) AS plus adjunct oAC vs. IV AS alone with regards to parasite clearance rate. This study will be conducted in African children, because they are the primary target population for such an intervention. Although the adequate standard-of-care treatment for UM is oral (PO) administration of an artemisinin-based combination therapy (ACT), we will treat participants with IV AS. Like ACT treatment of UM, AS is the WHO-recommended first-line treatment for SM (1). In order for the data obtained from UM cases to be meaningful for our future studies in children with SM, we will administer AS to the UM cases in this trial via the same IV route that is used to administer AS to SM cases. Exploratory objectives include: (i) to compare the kinetics of plasma cytokines in both groups, and (ii) to preserve RNA for gene transcription analysis for future studies into the mode of action of oAC. The study will be nested within an NIAID-funded study (Principal Investigators Drs. Fairhurst, Diakite) that assesses parasite clearance rates in response to AS treatment in Kenieroba (6). Children aged 2-10 years with UM and initial parasite densities 10,000 70,000 parasites per micro L will be enrolled. Parasite clearance rates will be expressed as the parasite half-life (Ph), estimated from parasite clearance curves using a formula that has been validated in this cohort (7). Children will be randomized 1:1 to receive IV AS+oAC or IV AS only, respectively, until complete specimen and data sets for 35 children per group are obtained. oAC will be administered as Actidose Aqua[registered] at 0, 6, 12, and 18 hours. AS will be administered IV following WHO recommendations for use of AS in SM (8), followed by 3 daily doses of amodiaquine (AQ). Subsequently and in a separate study, we plan a proof-of-concept RCT to determine whether adjunct oAC reduces disease severity and morbidity (assessed by scoring systems (9)) in hospitalized children with SM and to define the mode of action of oAC. Since oAC is a licensed, inexpensive drug without sophisticated storage requirements, which has an extremely long shelf life at room temperature and can be given orally or via nasogastric tube at high doses without major side effects (4, 10), this drug has an ideal profile for use at the primary health-care level to reduce mortality from SM, or even prevent the development of SM.

ELIGIBILITY:
* INCLUSION CRITERIA

  1. Age 2 to 10 years, inclusive
  2. Resident of Kenieroba
  3. Uncomplicated malaria*
  4. P. falciparum density 10,000 70,000/micro L, inclusive
  5. Willingness to participate in the study as evidenced by informed consent of the child s parent or guardian
  6. Ability to swallow oral medication

Uncomplicated malaria: axillary temperature >37.5oC or history of fever in the past few days and no criteria of SM (see next paragraph) and no other etiologies of febrile illness (e.g., respiratory tract infection) on clinical examination.

Severe P. falciparum malaria: parasitemia of any density and any one of the following: coma (Blantyre coma score less than or equal to 2), convulsions (witnessed by investigator), severe prostration, severe anemia (hemoglobin less than or equal to 6 g/dl), respiratory distress, hypoglycemia (serum glucose less than or equal to 40 mg/dl), jaundice/icterus, shock (systolic blood pressure less than or equal to 70 mmHg, rapid pulse, cool extremities), cessation of eating and drinking, repetitive vomiting.

EXCLUSION CRITERIA

1. Severe malaria
2. Any medical condition or history, including allergy to AS, AQ, artemether or lumefantrine, that poses a risk to the prospective participant
3. Any condition that in the opinion of the investigator would render the participant unable to comply with the protocol (e.g., psychiatric disease)
4. Any health condition that in the opinion of the investigator would confound data analysis or pose unnecessary risks to study participants (e.g., severe malnutrition, acquired or inherited immunodeficiency)
5. Requirement for any medication for any concurrent illness or condition
6. Participation on cohort study #13-I-N107
7. Repetitive vomiting

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2013-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rick M Fairhurst, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Universite des Sciencies, Techniques et Technologies de Bamako, Bamako, Mali

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AS + oAC: All children will receive Artesunate (AS) 2.4 mg/kg IV at 0 and 12 h, 24 h, and 48 h. Children in the AS+oAC group will be given weight-based doses of oAC (Actidose Aqua) (Table 1) at 0, 6, 12, and 18 h. All children will then receive amodiaquine.
  Actidose Aqua: Actidose Aqua (oAC, Paddock Laboratories) is sold over the counter in the US in bottles containing 25 g/120 mL (NDC # 0574-0121-04) or 50 g/240 mL (NDC # 0574-0121-08). oAC is stable at room temperature.
  Artesunate: Artesunate (AS) obtained from Guilin Pharma (Shanghai), the only pharmaceutical company GMP pre-qualified by the WHO. The product artesunate for injection + 5% sodium carbonate inj + 0.9% sodium chloride inj will be delivered in vials of 30 mg and 60- mg vials, respectively, and will be dosed at 2.4 mg/kg as recommended for SM treatment by the WHO
  Amodiaquine: Amodiaquine obtained from Pfizer (Dakar), is provided as 200-mg tablets or syrup (50 10 mg/mL), and will be provided as age-based doses.
Period: Overall Study
Arm/Group | AS + oAC | AS Only (Water)
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AS + oAC: All children in the AS+oAC group will receive artesunate (AS) 2.4 mg/kg IV at 0, 12, 24, and 48 h, and weight-based doses of oral activated charcoal (oAC; Actidose Aqua; according to Table 1) at 0, 6, 12, and 18 h. All children will then receive age-based doses of amodiaquine.
- AS Only (Water): All children in the AS Only group will receive artesunate (AS) 2.4 mg/kg IV at 0, 12, 24, and 48 h, and weight-based volumes of clean water at 0, 6, 12, and 18 h. All children will then receive age-based doses of amodiaquine.
- Total: Total of all reporting groups
Arm/Group | AS + oAC | AS Only (Water) | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.314 (2.166) | 5.600 (2.117) | 5.896 (2.168)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 18 | 38
  Male | 15 | 17 | 32
Weight [Mean (Standard Deviation); unit: Kilograms] | 19.29 (5.120) | 17.87 (4.568) | 18.59 (4.868)
Hemoglobin concentration [Mean (Standard Deviation); unit: grams per deciliter] | 10.93 (3.193) | 10.15 (1.047) | 10.54 (2.391)
Temperature [Mean (Standard Deviation); unit: degrees Celsius] | 36.37 (0.3511) | 36.45 (0.3988) | 36.41 (0.3751)
Parasite density [Mean (Standard Deviation); unit: log10(parasites per microliter)] | 4.421 (0.2569) | 4.459 (0.2592) | 4.440 (0.2569)

OUTCOME MEASURES:

1. Primary Outcome: Parasite Clearance Half-life
Description: To compare parasite clearance half-life in patients treated with IV AS + oAC or IV AS alone; parasite clearance half-life is the time it takes for the parasite density to decrease by half, and can be assessed by analysing frequent parasite density counts at 0, 2, 4, 6, 8, 12, 18, 24, 30, 36, 42, and 48 hours after initiating treatment.
Time Frame: During patient treatment
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | AS + oAC | AS Only (Water)
Number analyzed (Participants) | 35 | 35
Hours | 1.733 (0.7206) | 1.973 (0.6221)
Statistical Analysis 1: Comparison: AS + oAC vs AS Only (Water); Test type: Superiority; p > 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Safety
Description: To assess the safety of adjunct treatment with oAC; specifically, children were hospitalized while their vital signs were measured, IV site inspected, state of consciousness assessed, and selected symptoms (nausea, vomiting, diarrhea, constipation, abdominal pain, headache, and dizziness) surveyed at 0, 2, 4, 6, 8, and 12 hours, and then every 6 hours until 48 hours or until parasitemia became undetectable (one negative thick blood film), whichever was later.
Time Frame: During patient treatment up to 48 hours
Population: Children who received treatment per protocol
Measure: Count of Participants; unit: Participants
Groups:
- AS + oAC: All children will receive Artesunate (AS) 2.4 mg/kg IV at 0 and 12 h, 24 h, and 48 h. Children in the AS+oAC group will be given weight-based doses of oAC (Actidose Aqua) (Table 1) at 0, 6, 12, and 18 h. All children will then receive amodiaquine.
  Actidose Aqua: Actidose Aqua (oAC) (Paddock Laboratories is sold over the counter in the US in bottles containing 25 g/120 mL (NDC # 0574-0121-04) or 50 g/240 mL (NDC # 0574-0121-08). oAC is stable at room temperature.
  Artesunate: Artesunate (AS) obtained from Guilin Pharma (Shanghai), the only pharmaceutical company GMP pre-qualified by the WHO. The product artesunate for injection + 5% sodium carbonate inj + 0.9% sodium chloride inj will be delivered in vials of 30 mg and 60- mg vials, respectively, and will be dosed at 2.4 mg/kg as recommended for SM treatment by the WHO
  Amodiaquine: Amodiaquine obtained from Pfizer (Dakar), is provided as 200-mg tablets or syrup (50 10 mg/mL), and will be provided as age-based doses.
Arm/Group | AS + oAC | AS Only (Water)
Number analyzed (Participants) | 35 | 35
Participants | 35 | 35

ADVERSE EVENTS:
Time Frame: Up to 72 hours
Arm/Group | AS + oAC | AS Only (Water)
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 6/35 | 5/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AS + oAC (N=35) | AS Only (Water) (N=35)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-09-04): https://cdn.clinicaltrials.gov/large-docs/82/NCT01955382/Prot_SAP_000.pdf